CLINICAL TRIAL: NCT03570437
Title: A 3-Arm Randomised Phase II Evaluation of Cediranib in Combination With Weekly Paclitaxel or Olaparib Versus Weekly Paclitaxel Chemotherapy for Advanced Endometrial Carcinoma or for Disease Relapse Within 18 Months of Adjuvant Carboplatin-paclitaxel Chemotherapy.
Brief Title: Does Cediranib With Paclitaxel, or Cediranib and Olaparib, Treat Advanced Endometrial Cancer Better Than Paclitaxel?
Acronym: COPELIA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manchester (Other)
Collaborators: AstraZeneca (Industry); Cardiff University (Other)
Responsible Party: Principal Investigator, Prof Gordon Jayson, Professor of Medical Oncology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R120537; ESR-15-11357 (Other Grant/Funding Number: AstraZeneca); 17/SC/0536 (Other: HRA); 216069 (Other: IRAS); 2016-004617-28 (EudraCT Number); U1111-1197-9991 (Other: WHO UTN)
Record Dates: First submitted 2018-05-31; First posted 2018-06-27 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Carcinosarcoma; Endometrial Neoplasms
Keywords: Endometrial; Cancer; Paclitaxel; Cediranib; Olaparib
MeSH Terms: conditions — Carcinosarcoma; Endometrial Neoplasms; Neoplasms | interventions — Paclitaxel; cediranib; olaparib

STUDY DESIGN:
Intervention Model Description: Randomised, three-arm open-label trial with multi-arm-multi-stage (MAMS) design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Paclitaxel (Active Comparator): Paclitaxel 80 mg/m2 administered on days 1, 8 and 15 of a 28-day cycle for up to 6 cycles.
  Interventions: Drug: Paclitaxel
- Arm 2: Cediranib and paclitaxel (Experimental): Cediranib 20 mg once daily for 28 days given with weekly paclitaxel 80 mg/m2 administered on days 1, 8 and 15 of a 28-day cycle for up to 6 cycles. Participants with stable disease or better will be able to continue cediranib once daily until disease progression.
  Interventions: Drug: Paclitaxel; Drug: Cediranib
- Arm 3: Cediranib and olaparib (Experimental): Cediranib 20 mg once daily with olaparib 300 mg twice daily, continuously on a 28 day cycle for up to 6 cycles. Participants with stable disease or better will be able to continue with olaparib and cediranib until disease progression.
  Interventions: Drug: Cediranib; Drug: Olaparib

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m2 on three days in a 28 day cycle (with 6 cycles)
  Other Names: L01CD01
  Arms: Arm 1: Paclitaxel; Arm 2: Cediranib and paclitaxel
Drug: Cediranib — 20 mg per day
  Other Names: AZD2171; 288383-20-0
  Arms: Arm 2: Cediranib and paclitaxel; Arm 3: Cediranib and olaparib
Drug: Olaparib — Olaparib tablets, 300 mg twice-daily
  Other Names: AZD2281; Lynparza; L01XX46
  Arms: Arm 3: Cediranib and olaparib

SUMMARY:
The COPELIA trial is evaluating two new tablet medications in endometrial cancer for the first time. It will include 129 women aged 16 years or older with advanced endometrial cancer whose cancer has worsened after their initial chemotherapy treatment. Participants will be allocated at random to one of three groups:

1. The first group (Arm 1) will receive a standard (routine) treatment for patients with endometrial cancer known as paclitaxel. This is a chemotherapy drug that is routinely used to treat patients with different cancers including ovarian, breast, lung and endometrial cancer. Paclitaxel works by stopping the growth of cancer cells.
2. The second group (Arm 2) will receive the standard paclitaxel treatment once a week in addition to a new drug called cediranib. Cediranib is a tablet medication and works by blocking new blood vessel formation. Cediranib has been tested in women with endometrial cancer before but not alongside chemotherapy treatment.
3. The third group (Arm 3) will receive two new tablet medications, cediranib and olaparib. Olaparib works by preventing cancer cells repairing DNA effectively. The use of olaparib and cediranib together has been shown to be effective in a common type of ovarian cancer but has not been evaluated as a treatment for endometrial cancer before.

The main objectives of the COPELIA trial are to work out:

1. Whether the two new treatments, cediranib-paclitaxel (Arm 2) and cediranib-olaparib (Arm 3) are more effective at controlling endometrial cancer than standard paclitaxel chemotherapy (Arm 1)
2. Whether the two new treatments cause more or fewer side-effects than standard chemotherapy
3. How each of these treatments impact on the daily life of women receiving the treatment by asking trial participants to regularly complete quality of life questionnaires
4. Whether we can learn how these treatments work in women with endometrial cancer by taking some additional blood tests for research.

DETAILED DESCRIPTION:
COPELIA is a phase II, randomised, three-arm open-label trial which will recruit 129 women aged 16 years or older, with advanced endometrial cancer who require further treatment after their initial chemotherapy treatment. Potential participants will be recruited from the hospital setting.

Participants will be allocated to one of the following three trial arms on a 1:1:1 basis using centralised internet randomisation, stratified for prognostic factors:

Arm 1: (Control Arm): Paclitaxel 80 mg/m2 administered on days 1, 8 and 15 of a 28-day cycle for up to 6 cycles.

Arm 2: Cediranib 20 mg once daily for 28 days given with weekly paclitaxel 80 mg/m2 administered on days 1, 8 and 15 of a 28-day cycle for up to 6 cycles. Participants with stable disease, partial response or complete response at 6 months as determined by RECIST v1.1 will be eligible to continue treatment with single agent cediranib once daily until disease progression.

Arm 3: Cediranib 20 mg once daily with olaparib 300 mg twice daily, continuously on a 28 day cycle for up to 6 cycles. Participants with stable disease, partial response or complete response at 6 months as determined by RECIST v1.1 will be eligible to continue treatment with both olaparib and cediranib until disease progression.

Randomisation will be balanced for histological subtype and the number of chemotherapy regimens for metastatic disease.

Recruitment to the trial is expected to take 30 months. The total duration of the trial is expected to be 55 months. Participants will receive initial trial treatments for up to six months as long as they remain progression free. As mentioned above, participants in the experimental arms may continue treatment with cediranib/olaparib beyond the six months, and beyond the end of the trial, if they remain progression free. The trial will end once all participants have met at least one of the criteria: completed 12 months' follow-up (including treatment), withdrawn from follow-up, been lost to follow-up, experienced disease progression, or died. Participants consent for their medical notes to be reviewed at later dates if required to obtain data such as overall survival.

The trial has a multi-arm-multi-stage (MAMS) design. The appropriate sample size was calculated for this MAMS design, which allows one (or both) ineffective experimental arms to be dropped following a planned interim analysis after 60 participants have been assessed at three months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced or recurrent endometrial carcinoma or carcinosarcoma.
2. Aged >16 years.
3. All participants must have received at least one prior line of platinum-based chemotherapy (either in the adjuvant or recurrent disease setting). In addition, ONE of the following must apply:

   1. have disease recurrence/ progression within 18 months of completing adjuvant chemotherapy and have received no cytotoxic chemotherapy for recurrent/ progressive endometrial cancer.

      OR
   2. have received one or two prior lines of cytotoxic chemotherapy for recurrent/ progressive endometrial cancer (not counting adjuvant treatment).
4. Dose-dense weekly paclitaxel is an appropriate treatment option.
5. Ability to provide written informed consent that includes genetic research on tissue derived from biopsies and biomarker research. (If a participant declines to participate in optional exploratory genetic research or the optional biomarker research, there will be no penalty or loss of benefit to the participant. The participant will not be excluded from other aspects of the study).
6. Willing and able to comply with the trial visits and undergo treatment as scheduled.
7. ECOG Performance Status 0-1.
8. Life expectancy greater than 16 weeks.
9. Measurable disease by RECIST v1.1 including at least one not previously irradiated lesion that is ≥ 10 mm in the longest diameter (lymph nodes must have short axis ≥ 15 mm) as determined by CT.
10. Adequate haematological function: Hb ≥ 90.0 g/l with no requirement for blood transfusion in the last 28 days, neutrophils ≥ 1.5 x 109/l, platelets ≥ 100 x 109/l; coagulation: INR <1.4 (unless therapeutically anti-coagulated) and APPT ratio <1.4.
11. Adequate liver function: bilirubin ≤1.5 x ULN, transaminases ALT and AST ≤2.5x ULN. (AST or ALT <5x ULN allowed in the presence of parenchymal liver metastases.
12. Adequate renal function defined as calculated creatinine clearance using modified Wright or Cockcroft-Gault formula ≥ 51 ml/min or measured radioisotopic GFR ≥ 51ml/min.
13. Negative or trace proteinuria reading on urine dipstick. Patients with 1+ proteinuria on dipstick must have ≤1+ proteinuria on consecutive dipstick taken no less than 1 week later. Patients with ≥2+ proteinuria on dipstick must have 24 hour urinary protein excretion ≤1 g.
14. Adequately controlled thyroid function, with no symptoms of thyroid dysfunction.
15. Ability to swallow oral medication (tablets).
16. Willing to stop taking herbal supplements, and (if allocated to Arm 3) willing to not consume grapefruit or grapefruit juice, during the treatment period and for 30 days after end of trial treatment.

Exclusion criteria

1. Prior treatment with dose-dense weekly paclitaxel.
2. Uncontrolled brain metastases or seizures. A scan to confirm the absence of brain metastases is not required.
3. Known positivity for hepatitis B, hepatitis C or HIV due to the risk of transmitting the infection through blood or other body fluids and potential for reactivation during treatment.
4. Resting ECG with QTc > 470 ms on 2 or more time points within a 24 hour period or family history of long QT syndrome.
5. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is two weeks.
6. Concomitant use of known strong CYP3A inducers (eg.phenobarbital,enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
7. Pregnant or lactating. Pregnancy status in women of child bearing potential will be confirmed via a serum or urine pregnancy test prior to randomisation, monthly during the treatment period, and at the end of treatment assessment.
8. Of child bearing potential AND not willing to ensure they use effective contraception throughout the treatment period and for six months following the end of treatment. Acceptable methods of contraception are:

   i. true sexual abstinence (when this is in line with the preferred and usual lifestyle of the participant) ii. a combination of male condom plus one of:
   * vasectomised sexual partner, with participant assurance that partner received post-vasectomy confirmation of azoospermia
   * Tubal occlusion
   * Intrauterine device provided coils are copper-banded
   * Etonogestrel implants (eg, Implanon®, Norplant®)
   * Normal and low dose combined oral pills
   * Hormonal shot or injection (eg, Depo-Provera)
   * Intrauterine system device (eg, levonorgestrel-releasing intrauterine system -Mirena®)
   * Norelgestromin/ethinyl estradiol transdermal system
   * Intravaginal device (eg, ethinyl estradiol and etonogestrel)
   * Cerazette (desogestrel). Cerazette is currently the only highly efficacious progesterone based pill.
9. Side effects of previous treatments have not resolved to grade 1 or less, with the exception of alopecia that is considered related to cytotoxic chemotherapy.
10. Radiotherapy, chemotherapy, surgery or tumour embolisation within 28 days before the first dose of IMP.
11. Additional concurrent anti-cancer therapy.
12. Causes of malabsorption, e.g. uncontrolled diarrhoea or poorly controlled stoma.
13. Bowel obstruction, fistulae, impending fistulation seen on radiological imaging, or extensive rectosigmoid involvement by cancer.
14. Inadequately controlled hypertension, defined as ≥150/90 mmHg.
15. Prior or concurrent therapy with a PARP or VEGF inhibitor.
16. Known hypersensitivity to olaparib, cediranib or any of the excipients of the products.
17. Known hypersensitivity to paclitaxel that in the opinion of the investigator would prevent administration of a weekly paclitaxel regimen.
18. Exposure to an investigational agent within 30 days or 5 half-lives (whichever is the longer) prior to enrolment.
19. Considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
20. Myelodysplastic syndrome (MDS), acute myeloid leukaemia (AML) or features suggestive of MDS/AML.
21. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years.
22. Prior allogeneic bone marrow transplant or double umbilical cord blood transplantation.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 3 months
  Progression free survival rate at 3 months

SECONDARY OUTCOMES:
Radiological response rate | Assessed from CT scans up to and including the CT scan which shows disease progression, up to 6 months
  Radiological response rate assessed by RECIST v1.1
Median progression free survival (PFS) | From date of randomisation to date of investigator-assessed objective progression via RECIST v1.1 or death from any cause in the absence of progression, up to 42 months
  Time from date of randomisation to date of investigator-assessed objective progression via RECIST v1.1 or death from any cause in the absence of progression.
6-month progression free survival (PFS) | 6 months
  Proportion of participants free from investigator assessed objective disease progression by RECIST v1.1, or death from any cause, six months from the date of randomisation.
Toxicities | Up to 30 days after end of treatment
  Toxicities of any grade associated with each regimen as assessed by CTCAE version 4.03.
Median overall survival | From date of randomisation to date of death, up to 42 months
  Median time from date of randomisation to date of death
Quality of life using a questionnaire | Up to 30 days after end of treatment
  Quality of life measured using the EORTC QLQ-C30 tool and EN24 endometrial cancer-specific module.

OTHER OUTCOMES:
Angiogenesis-related cytokines | Up to 30 days after end of treatment
  Plasma concentration of circulating angiogenesis-related cytokines.
Circulating tumour cells (CTCs) | From randomisation until up to 30 days after end of treatment
  Proportion of participants with detectable CTCs at baseline, and the correlation between CTC levels and radiological response.
Gamma H2AX in circulating tumour cells | From randomisation until up to 30 days after end of treatment
  Evaluation of gamma H2AX in CTCs will be used as an exploratory tool to correlate presence or absence with radiological response.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Jayson, Principal Investigator — The Christie NHS Foundation Trust
Locations (15):
- United Kingdom (15):
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Royal Surrey County Hospital, Guildford, Surrey
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Bristol Haematology & Oncology Centre, University Hospitals Bristol NHS Foundation Trust, Bristol
  - Velindre Cancer Centre, Velindre University NHS Trust, Cardiff
  - Beatson West of Scotland Oncology Centre, Glasgow
  - Airedale NHS Foundation Trust, Keighley
  - Hope Clinical Trials Facility, Leicester Royal Infirmary, Leicester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - University College London Hospitals NHS Foundation Trust, London
  - Guys & St Thomas NHS Trust, London
  - Royal Marsden Hospitals, London
  - The Christie NHS Foundation Trust, Manchester
  - Northern Centre for Cancer Care, Freeman Hospital, Newcastle upon Tyne
  - The Churchill Hospital, Old Road, Headington, Oxford

IPD SHARING:
Plan to Share IPD: No